CLINICAL TRIAL: NCT01637194
Title: A Phase I Evaluation of Cetuximab and RAD001 in Patients With Solid Tumors
Brief Title: Cetuximab and Everolimus in Treating Patients With Metastatic or Recurrent Colon Cancer or Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 06-043; NCI-2011-02971 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-20; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Colon Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Stage IVA Colon Cancer; Stage IVA Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVA Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Colon Cancer; Stage IVB Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVB Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IVC Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Tongue Cancer
MeSH Terms: conditions — Colonic Neoplasms; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Everolimus; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor, monoclonal antibody therapy) (Experimental): Patients receive everolimus PO QD on days -14 and then 1-28. Patients also receive cetuximab IV over 60-120 minutes on days -7 and then once weekly beginning on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Biological: cetuximab; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of cetuximab when given together with everolimus in treating patients with metastatic or recurrent colon cancer or head and neck cancer. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of the tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Everolimus may stop the growth of tumor cells by blocking blood flow to the tumor. Giving cetuximab together with everolimus may be an effective treatment for colon cancer or head and neck cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety, dose-limiting toxicity and maximum tolerated dose of daily RAD001 (everolimus) when given in combination with a fixed dose of weekly cetuximab in patients with solid tumors.

SECONDARY OBJECTIVES:

I. Determine whether a pharmacokinetic interaction exists between RAD001 and CETUXIMAB in patients treated with this regimen.

II. Determine preliminary clinical evidence of anti-tumor activity by time to progression and Response Evaluation Criteria in Solid Tumors (RECIST) criteria with this regimen.

III. Determine the association between clinical outcomes and biologic markers that may predict sensitivity of a tumor in patients treated with this regimen.

IV. Determine the pharmacodynamic effects of this regimen on post-therapy tumor and/or skin specimens.

OUTLINE: This is a dose-escalation study of everolimus.

Patients receive everolimus orally (PO) once daily (QD) on days -14 and then 1-28. Patients also receive cetuximab intravenously (IV) over 60-120 minutes on days -7 and then once weekly beginning on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed advanced solid tumors
* Patients who are refractory to standard therapy; patients with metastatic, irinotecan-refractory colon cancer, or recurrent/metastatic head and neck cancer may enroll, as cetuximab monotherapy is among the standard options for such patients; patients with locally advanced, treatment-naïve head and neck cancer who are candidates for radiation with cetuximab are not eligible, as radiation provides them a survival benefit, and the number of projected cetuximab doses would be only seven
* Development of new lesions or an increase in preexisting lesions on bone scintigraphy, computed tomography (CT), magnetic resonance imaging (MRI) or by physical examination; patients in whom the sole criterion for progression is an increase in a biochemical marker, e.g., carcinoembryonic antigen (CEA), or an increase in symptoms, are not eligible
* No radiotherapy (unless palliative), treatment with cytotoxic agents, or treatment with biologic agents =< 3 weeks prior to registration on this study (6 weeks for mitomycin or nitrosoureas); >= 2 weeks must have elapsed from any prior surgery or hormonal therapy; patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment); patients with persisting, stable chronic toxicities from prior treatment =< grade 1 are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =<2 (Karnofsky >= 60%)
* Life expectancy of > 3 months
* Hemoglobin >= 9 g/dL
* Leukocytes >=3 K/mm^3
* Absolute neutrophil count >= 1.5 K/mm^3
* Platelets >= 100 K/mm^3
* Total bilirubin within institutional normal limits
* Hepatitis B panel negative
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN)
* Creatinine within 1.5 x ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; complete abstinence) prior to study entry and for the duration of study participation and for 3 months after the conclusion of study therapy, and must have a negative serum or urine pregnancy test =< 7 days prior to registration; pregnant and nursing patients are excluded because the side effects of the combination of cetuximab and RAD001 on a fetus or nursing child are unknown; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; sexually active men must also use appropriate contraception method and should not father a child while receiving therapy during this study
* Ability to understand and the willingness to sign a written informed consent document
* Fasting serum cholesterol < 350 mg/d L and triglycerides < 400 mg/d L
* Able and willing to undergo pharmacokinetic (PK) and pharmacodynamic (PD) testing as outlined in this protocol; if however the tumor is not amenable to the PD requirements of the protocol, the patient must be willing and able to undergo skin biopsy

Exclusion Criteria:

* Chronic treatment with systemic steroids or another immunosuppressive agent
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis or on therapeutic anticoagulation (except low dose coumadin)
* Patients may not have received prior cetuximab therapy
* Patients may not be receiving any other investigational agents; in addition, patients must not have received investigational treatment =< 30 days prior to registration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study
* Patients with chronic active hepatitis B or recent hepatitis B infection (hepatitis B surface antigen [HepB sAg] or immunoglobulin M [IgM] antibody to hepatitis B core antigen [IgM antiBc] positive) are ineligible because these patients are at increased risk of reactivation of the hepatitis B virus which may be fatal due to the immunosuppressive properties of RAD001
* Known human immunodeficiency virus (HIV)-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, oxygen dependent pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements; other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper gastrointestinal [GI] tract ulceration)
* All WOCBP MUST have a negative pregnancy test =< 7 days prior to registration; if the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | Day -14 through Day 28 of Cycle 1
  Dose-limiting toxicity defined as any grade 3 or greater non-hematologic, grade 4 thrombocytopenia, grade 4 neutropenia lasting more than 5 days, grade 4 febrile neutropenia requiring hospitalization or treatment delay more than 2 weeks due to unresolved toxicity.

SECONDARY OUTCOMES:
Composite Pharmacokinetic (PK) Analysis | At days -14, 1,and 22 at 1, 2, 3, 6, and 24 hours after drug treatment and day -7 and prior to dosing on day -4
  PKs derived from serum concentrations versus time for RAD001 on day -14, 1, and 22 at 1, 2, 3, 6, and 24 hours after drug administration as well as day -7 (h 168) and prior to dosing on Day 4.
Preliminary clinical evidence of anti-tumor activity by time to progression and RECIST criteria with this regimen | Baseline and every 2 courses (8 weeks)
Association between clinical outcomes and biologic markers that may predict sensitivity of a tumor in patients treated with this regimen | Baseline, 24 hours post-treatment on day 22
Pharmacodynamic effects of this regimen on post-therapy tumor and/or skin specimens | At baseline, 24 hours post-therapy on day 22

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burtness, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States